CLINICAL TRIAL: NCT01255007
Title: Prospective Comparison of 3T Gd-EOB-DTPA-enhanced MRI, Diffusion Weighted MR Imaging and MDCT of Colorectal Liver Metastases for Preoperative Detection and Assessment of Treatment Response Following Chemotherapy Treatment
Brief Title: Comparison of Primovist-enhanced MRI, Diffusion Weighted MRI and Multidetector CT of Colorectal Liver Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN100405CE2010
Record Dates: First submitted 2010-12-03; First posted 2010-12-07 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Colorectal Liver Metastases
Keywords: Colorectal; liver; metastases; Primovist; MRI; CT; cancer; resection; MDCT; Diffusion; Weighted; 3T
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; Body Weight | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Post chemotherapy group (Experimental): The first group consists of patients with colorectal liver metastases who have had treatment with chemotherapy and are now awaiting surgery. This group would have had Multidetector Liver CT (MDCT) imaging prior to the chemotherapy, and will now undergo post chemotherapy MDCT as part of standard clinical care in addition to Gd-EOB-DTPA enhanced liver MRI and Diffusion Weighted MRI (DW-MRI). The MRI will be performed as an additional imaging investigation after obtaining informed consent.
  Interventions: Other: MR imaging
- Pre and Post Chemotherapy Group (Experimental): The second group consists of patients with colorectal liver metastases who are due to receive neoadjuvant chemotherapy. This group will be imaged prior to receiving and after receiving chemotherapy. This will all be done prior to surgical resection of their colorectal liver metastases.
  Interventions: Other: MR imaging

INTERVENTIONS:
Other: MR imaging — Primovist enhanced MRI, Diffusion weighted MRI

SUMMARY:
1. Primovist-enhanced Magnetic resonance imaging (MRI) and Diffusion Weighted MRI (DW-MRI) is superior to Multidetector Computed axial Tomography (MDCT) in the detection of colorectal liver metastases. Fatty changes in the liver after chemotherapy treatment likely reduces the chances of seeing metastatic lesions on CT especially when the lesions are small (<10 mm). When compared with CT, Primovist-enhanced MRI and DW-MRI have the potential to provide higher contrast resolution enabling better detection of colorectal liver metastases following chemotherapy.
2. Primovist-enhanced MRI and DW-MRI are superior to CT in assessing and predicting treatment response of patients with colorectal liver metastases to chemotherapy. Primovist-enhanced MRI by providing superior resolution may provide improved accuracy in metastatic lesion margin detection thereby providing higher accuracy in estimating tumor response based on size criteria. DW-MRI provides information indirectly about tumor composition and therefore is likely to be superior to MD-CT in assessing treatment response.

Two groups of patients will be analyzed. The second group consists of patients with colorectal liver metastases who are to go for chemotherapy prior to surgery for metastases resection. This group will be CT and MRI scanned prior to chemotherapy and after chemotherapy. The first group of patients will consist of those patients who have already received chemotherapy and are likely to have surgery to resect liver metastases. This group will have only one set of scans done 4-6 weeks prior to their operation. The pathology of the resected metastases and CT and MRI images will be analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colorectal liver metastases already treated by chemotherapy and scheduled for surgical resection
* Patients with colorectal liver metastases scheduled to receive chemotherapy with possibility of future liver resection.

Exclusion Criteria:

* Acute or Chronic Renal Disease with Estimated GFR (eGFR) <30 mL/min.
* Hypersensitivity to MRI contrast or CT contrast or to any ingredient in the formulation or component of the container.
* Patients with: acute or chronic severe renal impairment (glomerular filtration rate <30 mL/min/1.73 m2), or acute renal insufficiency of any severity due to the hepato-renal syndrome or in the perioperative liver transplantation period.
* General contraindications to MRI such as pacemaker or ferromagnetic implants.
* Severe cardiovascular problems
* Pregnant or nursing women
* Age <18 years
* Liver Surgery is not a possibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-09; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To establish superiority of Primovist-enhanced liver MRI and DWI to MDCT in the preoperative detection of colorectal liver metastases in patients who have received prior chemotherapy by comparison against pathology or Intra-operative ultrasound. | 18 months

SECONDARY OUTCOMES:
To compare diagnostic performance of MDCT, Diffusion Weighted MR and Primovist-enhanced MRI in the differentiation of viable from non-viable metastatic tumour compared to reference standard of pathology. | 18 months
To investigate in the cohort of patients who have pre and post-chemotherapy MRI the role of DWI in predicting treatment response by baseline pretreatment Apparent Diffusion Coefficient (ADC) values. | 18 months
To assess performance of Primovist-enhanced MRI, DW-MRI and MDCT in assessment of treatment response following chemotherapy in the cohort of patients who have pre and post-chemotherapy MRI. | 18 months
To compare accuracies of Primovist-enhanced MRI and DWI to MDCT in the characterization of non-metastatic liver lesions against histopathology or intra-operative ultrasound. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Jhaveri, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada